CLINICAL TRIAL: NCT06928207
Title: A Randomized Experiment of Malaria Diagnostic Testing and Conditional Treatment Subsidies to Increase the Proportion of Malaria Patients Receiving an ACT
Brief Title: Private Medicine Retailer-based Trial of Malaria Tests and Conditional Treatment Subsidies Among Patients With Fever
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinton Health Access Initiative Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NHREC/01/01/2007- 19/05/2023
Record Dates: First submitted 2025-02-03; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-02

CONDITIONS: Malaria Falciparum
Keywords: Malaria; Private sector; Private Medicine Retailers; Drug shops; Subsidies; Case management; RDT; ACT; Nigeria
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Intervention Model Description: Private medicine retailers are recruited through a readiness assessment survey. A total of 60 licensed PMRs (based on a list provided by Pharmacy council Nigeria and NAPPMED) in the two targeted LGAs will be randomly selected and visited by trained data collectors and asked to participate in a short survey. The purpose of the survey is to determine (i) whether they are registered and (ii) willingness to participate in the study. Following the readiness assessment, a random sample of 24 PMRs are selected from eligible PMRs. Out of these 20 PMRs will be randomly selected for inclusion in the study with the remaining 4 PMRs serving as backups.
Who Masked: Outcomes Assessor
Masking Description: Primary outcome data is collected through Exit Interviewers. Exit interviews are conducted on randomly selected days each month and data collectors will be randomly assigned to participating private retailer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Free RDTs and conditional ACT subsidy: Patients visiting PMRs in this arm will receive a low-cost ACT if they use a low-cost RDT and have a positive test result.
  Interventions: Combination Product: Provide the diagnostic (RDT) for free to clients suspected of having malaria and provide a subsidized ACT to only those testing positive
- Control (No Intervention): Control: Standard practice

INTERVENTIONS:
Combination Product: Provide the diagnostic (RDT) for free to clients suspected of having malaria and provide a subsidized ACT to only those testing positive — To promote the use of the recommended first line drug, we implement a conditional subsidy. The retail provider is given the malaria diagnostic for free and is instructed to test clients suspected of having malaria. Only if the test is positive, the provider is instructed to provide the ACT at a low cost.
  Arms: Intervention arm

SUMMARY:
The goal of this study observational study is to test the effect of conditional subsidies for Rapid Diagnostic Tests (RDT) and Artemisinin Combination Therapies (ACT) on improving the management of malaria fevers that seek care in the retail sector. The main question it aims to answer is:

• Would a conditional subsidy scheme increase the proportion of clients with malaria receiving an ACT? Researchers will compare the proportion of patients with malaria receiving an ACT in the intervention arms to the control arm. Retail providers in the intervention arm have access to free RDTs and subsidized ACTs distributed by the research team and are asked to use a recommended retail price for the RDT and ACT. In addition, the providers in the intervention arm are trained in the use of RDTs and a mobile app that will prompt them to take and upload a picture of the RDT result. Retail providers in the control arm are trained in the use of RDTs but do not receive free RDTs or subsidized ACTs.

DETAILED DESCRIPTION:
The ultimate goal of the conditional subsidy scheme is to increase the proportion of patients with malaria that receives an artemisinin combination therapy (ACT) at the point of sale.

The objective of this study is to test the effect of providing low-cost malaria rapid diagnostic tests (RDT) and Artemisinin Combination Therapies (ACTs) to patients on improving the management of malaria fevers that receive care in private medicine retailers (PMR). During the study, malaria RDTs are provided free of charge to the private provider to conduct malaria-RDT testing at a low cost (at a set recommended retail price) for patients with a malaria-like illness. Subsidized ACTs are provided to the provider, conditional on the provider conducting the malaria RDT and selling the ACT at a low cost to patients testing positive for malaria. Outcomes will be measured by exit interviews on random days each month at participating PMRs.

ELIGIBILITY:
Inclusion Criteria:

* Participants who tested in the Private Medicine Retailer and/or purchased antimalarial (s) for themselves.
* Individuals with malaria-like illness must be present at recruitment.
* Older than one year of age.

Exclusion Criteria:

* Any individual with signs of severe illness requiring immediate referral.
* Individuals who have taken an antimalarial in the last seven days, including for the current illness.
* Patients <18 years without a parent or legal guardian present.
* Adults who are unable to consent for themselves

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-31 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
ACT uptake among patients testing positive for malaria during the exit interview | From enrollment exiting the PMR until the rapid test is conducted and the exit interview is concluded (approx 30 min)
  The proportion of patients with malaria that purchased an ACT during their visit to the PMR. For this outcome, a patient with malaria is anyone who has a malaria RDT performed and tests positive at the exit interview.

SECONDARY OUTCOMES:
Case management of patients visiting the PMR suspected of having malaria | From enrollment exiting the PMR until the rapid test is conducted and the exit interview is concluded (approximately 30 min)]
  The proportion of patients suspected of malaria cases that are managed appropriately (tested for malaria in the PMR or elsewhere but with proof and purchase any ACT following a positive RDT test result or do not purchase an ACT after a negative RDT rest result)
Out of pocket expenses incurred by patients suspected of having malaria | From enrollment exiting the PMR until the rapid test is conducted and the exit interview is concluded (approximately 30 min)]
  The out-of-pocket expenses incurred in the PMR by patients suspected of having malaria for ACTs and RDTs
Proportion of untested clients who purchase ACTs | From enrollment exiting the PMR until the rapid test is conducted and the exit interview is concluded (approx 30 min)
  Proportion of clients visiting the PMR that did not test in the drugshop and purchased ACTs

CONTACTS AND LOCATIONS:
Locations (1):
- Private Medicine Retailers, Igabi and Kajuru LGA, Kaduna State, Nigeria

IPD SHARING:
Plan to Share IPD: No